CLINICAL TRIAL: NCT06672653
Title: PREPAP Study: Tolerance and Effectiveness of the Monoterpenoid Zinc Tetra-ascorbo-camphorate (C14) on the Genital Load of Oncogenic HPV (HR-HPV) and Precancerous Cervical Lesions: Research With Direct Individual Benefit
Brief Title: Tolerance and Effectiveness of C14 on HPV Infection
Acronym: PREPAP
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MGB Pharma (Industry)
Responsible Party: Principal Investigator, Serge Tonen-Wolyec, Infectiologist, MD, PhD; Academic General Secretary of the University of Bunia; Member of the Société Africaine sur le SIDA (SAA) and Société Française de Microbiologie (SFM)., University of Kinshasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PREPAP/CER/006/GEAK/2024
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: HPV-induced Cancers; HPV Infections; HIV; Cervical Cancers; Trial; C14; Monoterpenoid Zinc Tetra-ascorbo-camphorate
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — Carbon-14

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C14 arm (Experimental): In this arm, particpants will received by vaginal syringe, 5ml of 1% C14, twice a day for 7 days, starting the first cure during the follicular phase of the cycle, just after the last menstrual period (S1), the second cure the following month (S5), the third cure 4 weeks later (S9) and the last cure 8 weeks later (S13).
  Interventions: Drug: The monoterpenoid zinc tetra-ascorbo-camphorate ("C14")
- Control arm (Placebo Comparator): In this arm, particpants will received by vaginal syringe, 5ml of distilled water, twice a day for 7 days, starting the first cure during the follicular phase of the cycle, just after the last menstrual period (S1), the second cure the following month (S5), the third cure 4 weeks later (S9) and the last cure 8 weeks later (S13).
  Interventions: Drug: Distilled water group

INTERVENTIONS:
Drug: The monoterpenoid zinc tetra-ascorbo-camphorate ("C14") — The trial phase will consist of hospital administration by vaginal syringe of 5ml of 1% C14, twice a day for 7 days, starting the first cure during the follicular phase of the cycle, just after the last menstrual period (S1), the second cure the following month (S5), the third cure 4 weeks later (S9) and the last cure 8 weeks later (S13). Gynaecological follow-up with HPV molecular testing and cervical smear will be performed two days after each course of treatment at S2, S6, S10, S14 and 2 weeks after the last course of treatment (S16). Unprotected sexual intercourse will not be permitted during each course of treatment, and for at least 72 hours before each genital swab.
  Arms: C14 arm
Drug: Distilled water group — Instead of C14, distilled water will be administered in this group.
  Arms: Control arm

SUMMARY:
The zinc monoterpenoid tetra-ascorbo-camphorate possesses broad-spectrum anti-viral properties in vitro, particularly against HIV, HSV and HPV. Its C14 formulation could be a promising candidate for in vivo clinical evaluation as a potential microbicide or therapeutic drug.

The aim of this clinical trial is to determine whether C14 is effective in reducing the genital viral load of HR-HPV and in treating low-grade dysplastic lesions of the cervix. It will also determine the tolerability of C14. The main questions to be answered by the clinical trial are as follows:

Does C14 reduce the genital HR-HPV viral load in participants with persistent HR-HPV infections? What medical problems do participants experience when taking C14? Researchers will compare C14 to a placebo (a similar substance that contains no drug) to see if C14 is effective in reducing genital C14 viral load and in treating low-grade dysplastic lesions of the cervix.

Participants will

receive four monthly treatments (5ml of C14 dissolved in distilled water administered twice daily [morning and evening] for seven days via vaginal syringe during the follicular phase) of C14 or placebo for 4 months and visit the clinic once every 2 weeks for examinations and tests. They will keep a diary of their symptoms and the number of times they keep the hospital appointment.

DETAILED DESCRIPTION:
1. Rationnal :

   The human papillomavirus (HPV) group includes 200 known viruses. Persistent high-risk HPV infection can cause cervical cancer, and is associated with cancers of the vulva, vagina, mouth/throat, penis and anus. Effective preventive interventions against HR-HPV exist in developed countries, such as the Gardasil and Cervarix vaccines. These interventions are implemented with great disparity in sub-Saharan Africa, where many African women carry high cervical viral loads of HR-HPV and precancerous and dysplastic lesions. The use of antimicrobial molecules would appear to be one way of improving the management of these women.

   The monoterpenoid zinc tetra-ascorbo-camphorate ("C14") thus possesses pleiotropic antimicrobial properties. Several in vitro experiments have demonstrated C14's viricidal activity against HIV (Shattock, 1997; Barré-Sinoussi, 2008) and HPV (Mboumba Bouassa, 2021). A phase I/II clinical trial of C14's tolerance-efficacy on genital oncogenic HPV load (HR-HPV) and on precancerous cervical lesions is now envisaged, with a view to boosting the development of C14 through a larger-scale trial.
2. Objectives

   2.1. General objective

   This research aims to contribute to the reduction of cervical cancer morbimortality through the in vivo evaluation of C14 as a potential microbicide or therapeutic drug against oncogenic HPV.

   2.2. Specific objectives :
   * Determine whether C14 is effective in reducing the genital viral load of HR-HPV and in treating low-grade dysplastic lesions of the cervix;
   * Evaluate the tolerability of C14 among volunteers.
3. Methods

3.1. Study design

The present study is a double-blind randomized placebo-controlled clinical trial. It will include 66 patients in Polyclinique Citadelle, a health centre in Bunia, Democratic Republic of the Congo. It is estimated to last 18 weeks considering final data collection for primary outcome measurements.

3.2. Participants

1. Inclusion criteria:

   The targeted population is all sexually-active women, aged at least 30 years old and who will give their informed consent to participate in the study.

   The reason for this target population is based on the natural history of HPV infection. HPV is acquired at the onset of sexual activity which occurs at around 15 to 20 years of age. Its prevalence is very high at a younger age and is often transient because most women will spontaneously eliminate the virus after some years. When it persists, HPV infection can take in average 10 years to lead to cervical cancer. Thus, testing is projected to start 10 years later after sexual debut in this case at 25 to 30 years old onward.
2. Exclusion Criteria:

Pregnant, breastfeeding and post-partum women will not be accepted in the study. In case of suspected or diagnosed cervical cancer, the women will be referred in a tertiary hospital for the proper management. Other exclusion criteria include: previous cervical surgery, medical history of any severe diseases, intake or application of other antivirals, known or suspected allergic or adverse response to the investigational product or its components and women who are unable to follow the study protocol.

3.3. Randomization procedures

Participants will randomize at a ratio of 1:1 through block randomization. Eligible participants were randomly assigned to one of two self-testing groups, C14 group or placebo-group, using sequentially numbered sealed randomization envelopes.

3.4. Procedures and follow-up

Before the start of the study, basic training will be organized for the doctors and nurses involved in the survey. This training will cover Good Clinical Practice (GCP), sample collection using the vaginal veil (V-V-Veil Up) and Thinprep cytobrushes, as well as procedures for Visual Inspection after application of acetic acid (VIA) and cryotherapy.

The preliminary phase of the trial will involve prospective recruitment of at least 420 women who meet our criteria. Formal informed consent will be obtained, and education on the importance of cervical cancer diagnosis and prevention with early treatment of possible pre-cancerous cervical lesions will be provided. Eligible volunteers will be invited to participate in a community-based cervical cancer screening program (VIA). Then, primary molecular screening for HR-HPV will be performed using a medical device for self-sampling of cervicovaginal secretions (Vaginal Veil Collector V-Veil Up UP2™, VVeil-Up Production SRL, Romania). Cervical vaginal secretions will be deposited in CytAll transport medium prior to PCR analysis using the Singu 20 extractor (Singuway, Shenzhen, China) and QuantGene 9600 thermocycler (Bioer Technology, Hangzhou, China). In case of presence of at least one HR-HPV (positive HPV test with Ct < 33), eligible participants will lie in lithotomy position on the gynecological table. After exposing the cervix with a speculum inserted into the vagina, the physician will take a cervical sample using Thinprep PreservCyt® solution (Hologic, Marlborough, USA) for cervical cytological analysis. Cervical lesions will be interpreted according to the Bethesda classification.

The trial phase will consist of hospital administration by vaginal syringe of 5ml of 1% C14, twice a day for 7 days, starting the first cure during the follicular phase of the cycle, just after the last menstrual period (S1), the second cure the following month (S5), the third cure 4 weeks later (S9) and the last cure 8 weeks later (S13). Gynaecological follow-up with HPV molecular testing and cervical smear will be performed two days after each course of treatment at S2, S6, S10, S14 and 2 weeks after the last course of treatment (S16). Unprotected sexual intercourse will not be permitted during each course of treatment, and for at least 72 hours before each genital swab.

The Phase I trial will be a tolerance test after the first course of treatment. All participants will complete the WHO clinical tolerance grid questionnaire during a medical examination. Physical and colposcopic examinations will be carried out, followed by an assay of pro-inflammatory, systemic and cervico-vaginal markers, and a hematological, hepatic and renal check-up.

The Phase II trial will be an efficacy trial after each course of treatment (four courses), comparing the efficacy of C14 between the two study arms. End-points will be virological (genital HR-HPV load) and cytological. Cytological controls will be carried out after 6 months and one year from the start of the trial.

3.5. Statistical analyses

Data will be collected in Excel data base using le Kobo collect KoboCollect software and the analyses will be performed with SPSS 20.0 (IBM, Atlanta, USA). Proportions will be compared using the x2 or Fisher's exact tests (when required). Student's t-test will be used for continuous variables. A Mc Nemar test will be used for within-patient comparisons where approriate. Nonnormally distributed variables will be transformed, or nonparametric tests (Wilcoxon or Kruskal-Wallis) will be used. Stepwise multivariate analyses will be performed, and all possible interactions up to order 2 will be tested. All reported P values will be 2-sided. For all statistical analyses a P value of ≤0.05 will be considered as statistically significant.

3..6. Ethical issues The PREPAP study is approved by the Institutional Ethical Committees of both the University of Kisangani and the Univwersity of Bunia. It will be conducted in full agreement with the principles of the "Declaration of Helsinki" and subsequent relevant amendments. All participants will provide written informed consent before entering the trial.

ELIGIBILITY:
Inclusion Criteria:

* sexually-active women
* aged at least 30 years old
* who will give their informed consent to participate in the study.

Exclusion Criteria:

* Pregnant
* breastfeeding and post-partum women will not be accepted in the study.
* previous cervical surgery, medical history of any severe diseases, intake or application of other antivirals
* known or suspected allergic or adverse response to the investigational product or its components
* women who are unable to follow the study protocol.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
genital HR-HPV load | From enrollment to the end of treatment at 16 weeks

SECONDARY OUTCOMES:
Virological cytological | From enrollment to the end of treatment at 16 weeks
  The aim here will be to verify whether C14 could cure low-grade cervical lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Polyclinique Citadelle, Bunia, Ituri, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saidi H, Jenabian MA, Gombert B, Charpentier C, Mannarini A, Belec L. Pre-clinical development as microbicide of zinc tetra-ascorbo-camphorate, a novel terpenoid derivative: potent in vitro inhibitory activity against both R5- and X4-tropic HIV-1 strains without significant in vivo mucosal toxicity. AIDS Res Ther. 2008 Jun 3;5:10. doi: 10.1186/1742-6405-5-10. PMID 18522743
- [Background] Mutombo AB, Tozin R, Simoens C, Lisbeth R, Bogers J, Van Geertruyden JP, Jacquemyn Y. Efficacy of antiviral drug AV2 in the treatment of human papillomavirus-associated precancerous lesions of the uterine cervix: A randomized placebo-controlled clinical trial in Kinshasa, DR Congo. (KINVAV study). Contemp Clin Trials Commun. 2017 Sep 28;8:135-139. doi: 10.1016/j.conctc.2017.09.008. eCollection 2017 Dec. PMID 29696202
- [Background] Mboumba Bouassa RS, Gombert B, Mwande-Maguene G, Mannarini A, Belec L. In vitro inhibitory activity against HPV of the monoterpenoid zinc tetra-ascorbo-camphorate. Heliyon. 2021 Jun 6;7(6):e07232. doi: 10.1016/j.heliyon.2021.e07232. eCollection 2021 Jun. PMID 34159277
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34159277/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29696202/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/18522743/